CLINICAL TRIAL: NCT02872948
Title: Diagnosis Accuracy of Noninvasive Screening by PCR Digital for Down Syndrom
Acronym: DIgiT21
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC14.185
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Trisomy 21
Keywords: Non invasive prenatal testing; Down Syndrome; Digital PCR
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — It is DNA samples of 100 pregnancies including 70 euploïdes foeti and 30 trisomies 21, the diagnosis of which will beforehand have been made by the foetal karyotype.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 70 euploïdes foeti samples: Patients with foetus euploïde ("no sick")
  Interventions: Genetic: Diagnostic
- 30 trisomies 21 samples: Patients with foetus reached(affected) by trisomy 21 ("sick")
  Interventions: Genetic: Diagnostic

INTERVENTIONS:
Genetic: Diagnostic

SUMMARY:
The main objective of this study is to estimate the intrinsic diagnostic qualities of the digital dPCR in the screening of T21 from a multicentrique sample of patients with pregnancies at high risk of T21 (risk > 1/250).

The profit expected from this technique is to propose to the encircled women a screening more successful than that of the screening combined(organized) of the 1st quarter, simple of realization and in a moderate cost. We thus propose here an original alternative(alternate) method to the exclusive, expensive and binding techniques of top-debit(-flow). The recent technical improvements and his(her,its) advantages medical - economic allow to envisage a reliable, strong and long-lasting use of the dPCR in clinical routine in the DPNI of T21 in most of the laboratories. This pilot project could serve for the later development of a study of clinical validation multicentrique of large scale(big turntable ladder).

DETAILED DESCRIPTION:
Context

Currently, non-invasive screening test for trisomy 21 (Down syndrome) is proposed to every pregnant woman. This first trimester combined test consists of ultrasound nuchal translucency measurement, associated with different maternal serum biochemical assay and maternal age.

Since the discovery of the presence of cell-free fetal DNA in maternal plasma, the noninvasive prenatal testing (NIPT), using mainly a massive parallel sequencing (MPS) approach, has been introduced. The chromosomal origin of each sequenced plasma DNA molecule and the over- or under-representation of any chromosome can be identified by MPS in maternal plasma. The specificity and sensibility of such high-throughput techniques are excellent, close to 100 %. However, MPS remains time-consuming, very expensive (> 1000 euros per patient) and can't be used in clinical routine in most genetics laboratories worldwide.

Digital PCR represents an interesting alternative to the MPS due to its targeted approach, cost (>10x less than MPS), speed and relative simplicity allowing a clinical routine practice. However, its clinical an analytical relevance remains insufficiently demonstrated in literature data . Therefore, our main objective is to evaluate the diagnosis accuracy of noninvasive screening by PCR digital for Down syndrome.

Expected results This study will assess the sensitivity, specificity and likelihood ratio with a satisfactory accuracy. The no call rate will be also evaluated and considered as a positive test.

The optimal number of replicates (leading to a false positive rate <5%) will be determined using a ROC curve. Our hypothesis is that the sensitivity of the screening test will be upper to 95% with a false positive rate <5%.

If results are conclusive, this pilot project will be a strong argument in favor of the development of a further large scale study. It may challenge current screening strategy and allow to propose an inexpensive, fast, and accessible NIPT of trisomy 21 to a large number of laboratories in our territory.

Experimental design We will evaluate this approach on a pregnant women cohort with high risk for T21 (>1/250), prospectively recruited from three regional hospitals with a cytogenetics laboratory. We propose to preform single-blind retrospective analyses of cell free DNA of 100 pregnancies (including 70 euploid and 30 T21fetuses). Results obtained with the dPCR approach will be compared with the fetal karyotype beforehand performed. Digital PCR analyses will be performed at the Grenoble University Hospital, our team having a significant experience in digital PCR technology. Digital PCR reactions will be done on a QuantStudio™ 3D (LifeTechnologies) with the commercial high density chips etched with 20,000 consistently-sized nanoscale reaction wells. To improve the analytical sensitivity, 10 replicates will be performed for each patient.

ELIGIBILITY:
Inclusion Criteria:

* major Patients
* unique(only) Pregnancies
* Screening combined(organized) by the 1st quarter of the trisomy 21 with risk > 1/250
* Patients wishing to realize a foetal taking with diagnostic aim
* Sent in maternity(maternity hospital) for this taking between 12 and 17 weeks of amenorrhea

Exclusion Criteria:

* Patient refusing to participate
* no Patient beneficiary of the Social Security or other diet
* Private person of freedom

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Sample multicentrique of patients with pregnancies at high risk of T21 (risk > 1/250)
Sampling Method: Probability Sample
Enrollment: 1260 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Intrinsic diagnostic qualities of the digital dPCR in the screening of T21 from a sample multicentrique of patients with pregnancies at high risk of T21 (risk > 1/250) | 24 months
  The main criterion is the estimation of the intrinsic qualities of the dPCR in the screening of T21. The sensibility of the screening will be favored and the reserved value will be the one giving a rate of acceptable positive forgery fixed to 5 %.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital center, Grenoble, France

REFERENCES:
- [Background] Cans C, Amblard F, Devillard F, Pison H, Jalbert P, Jouk PS. Population screening for aneuploidy using maternal age and ultrasound. Prenat Diagn. 1998 Jul;18(7):683-92. PMID 9706649
- [Result] Coutton C, Abada F, Karaouzene T, Sanlaville D, Satre V, Lunardi J, Jouk PS, Arnoult C, Thierry-Mieg N, Ray PF. Fine characterisation of a recombination hotspot at the DPY19L2 locus and resolution of the paradoxical excess of duplications over deletions in the general population. PLoS Genet. 2013 Mar;9(3):e1003363. doi: 10.1371/journal.pgen.1003363. Epub 2013 Mar 21. PMID 23555282
- [Result] Nadeau G, Coutton C, Amblard F, Michalowicz G, Frasca S, Fertin A, Devillard F, Satre V, Usson Y, Jouk PS. Interphase fluorescent in situ hybridization detection of the 7q11.23 chromosomal inversion in a clinical laboratory: automated versus manual scoring. Clin Chem Lab Med. 2013 Apr;51(4):e41-4. doi: 10.1515/cclm-2012-0416. No abstract available. PMID 23072851
- [Result] Coutton C, Bidart M, Rendu J, Devillard F, Vieville G, Amblard F, Lopez G, Jouk PS, Satre V. 190-kb duplication in 1p36.11 including PIGV and ARID1A genes in a girl with intellectual disability and hexadactyly. Clin Genet. 2013 Dec;84(6):596-9. doi: 10.1111/cge.12113. Epub 2013 Mar 25. No abstract available. PMID 23521658
- [Result] Ben Khelifa M, Coutton C, Zouari R, Karaouzene T, Rendu J, Bidart M, Yassine S, Pierre V, Delaroche J, Hennebicq S, Grunwald D, Escalier D, Pernet-Gallay K, Jouk PS, Thierry-Mieg N, Toure A, Arnoult C, Ray PF. Mutations in DNAH1, which encodes an inner arm heavy chain dynein, lead to male infertility from multiple morphological abnormalities of the sperm flagella. Am J Hum Genet. 2014 Jan 2;94(1):95-104. doi: 10.1016/j.ajhg.2013.11.017. Epub 2013 Dec 19. PMID 24360805